CLINICAL TRIAL: NCT02451085
Title: The Effect of a Telerehabilitaion Program on Gait and Balance in Patients After Hip Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reuth Rehabilitation Hospital (Other)
Collaborators: Video Therapy Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-2
Record Dates: First submitted 2015-04-20; First posted 2015-05-21 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis, Hip; Hip Injuries
Keywords: hip; surgery; Replacement
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- remote rehabilitation group (Experimental): 'training with video therapy' a domestic exercise plan through remote rehabilitation system based on short film. (http://videotherapy.co/vt/home.php), the plan will include installation of exercises adapted according to the physical condition of the patient. The content of each exercise is dynamic and variable. The difference between each exercise and the other depends on the feedback that the patient fills at the end of each exercise and sends to the therapist. Before each exercise, it is shown with explanations about the importance of performing it the way of performing. Furthermore, during the training, the patient listens to vocal explanation about the quality and importance of performing the exercise, and a vocal counting is heard and then a positive feedback is given.
  Interventions: Behavioral: training with video therapy
- conventional exercise group (Other): will receive instruction for self-training as accepted today through exercise sheet. The exercises will be suited to the ones provided to the patients in the intervention group. Moreover, a follow-up sheet will be given to the patients to fill in order to receive a feedback at the end of experiment. The training duration will be identical in both groups and will last for 30-45 minutes, three times a week.
  Interventions: Behavioral: conventional exercise

INTERVENTIONS:
Behavioral: training with video therapy — training with video therapy
  Arms: remote rehabilitation group
Behavioral: conventional exercise — training in conventional way
  Arms: conventional exercise group

SUMMARY:
The purpose of the present study is to examine whether an intervention plan based on exercise through remote rehabilitation system leads to improvement in characteristics of walking and balance among patients after hip replacement surgery compared to the current conventional way of exercise among these patients.

DETAILED DESCRIPTION:
Osteoarthritis is the main and most common reason for replacing hip joint and in forecast for 2020s this will be the fourth reason that causes disabilities throughout the world. Osteoarthritis causes not only physical limitation but also damage to the quality of life. Pain and functional limitation appear among about 10% of men and 18% of women over the age of 60. Pain and limitation in range of movement, functional decrease in daily functioning such as walking distance and endurance, difficulty in climbing up and down stairs are typical signs among those patients before surgery and treatment.

Other physical defects following hip replacement surgery last for over a year and they include a decrease in muscle strength round the operated hip, a defect in keeping balance in the operated leg and a functional decrease that includes decrease in walking speed, damage in the ability of climbing up and down stairs and difficulty in standing up.

Physical rehabilitation has importance among patients after hip joint surgery. Rehabilitation begins on the first stage at the rehabilitation hospital and continues after discharge at the community, at home or at the clinic. Often, the need for a continuing rehabilitation treatment after discharge exceeds the treatment provided actually by healthcare in Israel because of various reasons e.g. residence in remote areas, loads of patients who need treatment and high costs of manpower and reaching the treatments.

Remote Therapy is an alternative means to the present therapy in clinics which is provided at the patient's home and thus solving these problems. Remote Therapy employs technological communication and thus enables the patient to continue the rehabilitation process independently with no need for reaching the clinic which makes it easier for the patient and saves economic costs for the financial agent.

The purpose of the present study is to examine whether an intervention plan based on exercise through remote rehabilitation system leads to improvement in characteristics of walking and balance among patients after hip replacement surgery compared to the current conventional way of exercise among these patients

ELIGIBILITY:
Inclusion Criteria:

* One to three months after hip surgery
* Age 50-85

Exclusion Criteria:

* Individuals with central neurological disability
* Dependent individuals in passing from bed to wheelchair
* Significant cognitive disability according to the attendant physician
* Individuals with vascular-based pathologies

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
GAITMAT | Base line; change after 6 weeks treatment; and change after 10 weeks
  is an electronic path used to measure the time (timing) and space via pressure sensors placed on a track. The purpose of the system is to measure the events that occur during movement, data on time and space is measured and walking speed
SMART STEP | Base line; change after 6 weeks treatment; and change after 10 weeks
  is an instrument which provides feedback during walking about the amount of burden that the patient places on his leg. A feedback about placing the burden on the whole foot, toes or on the heel is possible. Investigators will set the minimal and maximal weight that we want the patient to reach while stepping. When the patient reaches the minimal weight, he will hear a single pip and when he reaches the maximal weight or more, he will hear two pips. In other words, this instrument gives us an indication for the patient's carrying of the weight- how much weight he placed on the leg while walking on each area and indication for the duration of the foot placed on the ground and in the air
BBS (Berg Balance Scale) | Base line; change after 6 weeks treatment; and change after 10 weeks
  the test includes 14 static and dynamic tasks for keeping balance. Each task receives a score from 0 to 4 points- according to the quality of task and performance time, maximal score of 56 points. Instructions regarding performing each task separately and the score of each task appear in the test form.
  The low performance in each task is considered in the score. In most tasks the patient is asked to keep a specific pose for a while. The score must be decreased if the patient does not meet the requirements of wished time or distance or if he gets external support or assisted by the tester.

SECONDARY OUTCOMES:
TUGT (Times Up And Go): | Base line; change after 6 weeks treatment; and change after 10 weeks
  A balance test which is measures by time, the ability of standing up from sitting position, walking for three meters, turning around and sitting down. This test examines the ability to integrate balance and movement including establishing movement, initiation, performing and completing a set of attached movements that we encounter in daily functioning.
THE FIVE SIT-TO-STAND TEST | Base line; change after 6 weeks treatment; and change after 10 weeks
  a physical test that integrates dynamic balance test. In this test the patient is asked to stand up and sit down five times continuously as quickly as possible on a standard chair and the tester measures the time.
MLEFS- LOWER EXTREMITY FUNCTIONAL SCALE | Base line; change after 6 weeks treatment; and change after 10 weeks
  subjective questionnaire that will assess their independency degree according to the subjective report of each patient. Result of 80/80 indicates full independency while 0/80 indicates external difficulty or disability in functioning
responsiveness to the treatment | 6 weeks
  At the end of each week a form is delivered to the patients in order to examine the responsiveness to the treatment; the form includes two questions regarding the performance of exercise. At the beginning of the experiment each patient receives a form and at the end of each week they must answer both questions and send the answers via SMS to the secondary investigator, or via fax.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jeaques Vatine, Prof, Principal Investigator — Reuth Rehabilitation Hospital; Alon Kalron, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Reuth Rehabilitation Hospital, Tel Aviv, Israel